CLINICAL TRIAL: NCT06928350
Title: Normal Values of Ambulatory 24-hour Oesophageal pH-impedance Monitoring in an Indian Cohort of Participants
Status: Recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: Oesophageal PH-01
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
Keywords: 24- hour pH impedance monitoring; GERD; Acid exposure; Healthy volunteers; Indian cohort; reflux episodes
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A group of 50 healthy volunteers: A sample size of 50 healthy volunteers will be enrolled

SUMMARY:
This study aims to determine normal 24-hour pH-impedance monitoring values, including acid exposure time (AET), in healthy Indian adults. It will help improve GERD diagnosis in India by providing population-specific data. The study will also explore how diet, body position, and nighttime reflux affect acid exposure. Healthy volunteers aged 18 and above will be monitored for 24 hours.

DETAILED DESCRIPTION:
This prospective study aims to establish normal 24-hour ambulatory pH-impedance monitoring values, including acid exposure time (AET), in healthy Indian volunteers. With an estimated GERD prevalence of 8-10% in India, current diagnostic criteria, such as the Lyon Consensus cut-off of 6%, may not be suitable for the Indian population due to differences in AET. The study will investigate the normative values of AET in healthy individuals and examine how factors such as diet, body position, and nocturnal reflux influence acid exposure and reflux episodes. By determining these standard values, the study seeks to enhance the accuracy of GERD diagnosis in India and improve understanding of reflux patterns specific to the Indian population. Participants will be healthy adults aged 18 and above, without gastrointestinal symptoms or major systemic diseases. The study will be conducted as a single-centre, 24-hour monitoring protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-50 years of age
* No gastro-intestinal symptoms
* No past GI or thoracic or spine surgery
* Not on any medications
* No history of recent alcohol intake (0 drinks in the past 1 month)
* Non smoker
* Normal BMI (18.5-22.9)

Exclusion Criteria:

* Any diagnosed systemic or organ specific disease (liver/kidney/heart/neurological disease, DM/HTN/Thyroid disease/ connective tissue disorder/inflammatory bowel disease/ irritable bowel syndrome)
* GERD symptoms/ functional dyspepsia
* Pregnant women or breast-feeding women
* Helicobacter pylori infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Normal values of ambulatory 24-hour oesophageal pH-impedance monitoring in an Indian cohort of healthy volunteers | The primary outcome measures include the percentage of time the esophageal pH is below 4 (acid exposure time) and the total number of reflux episodes detected by impedance monitoring in both proximal and distal channels, assessed over a 24-hour monitorin
  The primary outcome measures include the percentage of time the esophageal pH is below 4 (acid exposure time) and the total number of reflux episodes detected by impedance monitoring in both proximal and distal channels, assessed over a 24-hour monitoring period.

CONTACTS AND LOCATIONS:
Locations (1):
- AIG hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim SY, Jung HK, Lee HA. Normal acid exposure time in esophageal pH monitoring in Asian and Western populations: A systematic review and meta-analysis. Neurogastroenterol Motil. 2021 Apr;33(4):e14029. doi: 10.1111/nmo.14029. Epub 2020 Dec 30. PMID 33377596
- [Result] Ramu B, Mohan P, Rajasekaran MS, Jayanthi V. Prevalence and risk factors for gastroesophageal reflux in pregnancy. Indian J Gastroenterol. 2011 May;30(3):144-7. doi: 10.1007/s12664-010-0067-3. Epub 2010 Dec 2. PMID 21125366
- [Result] Zhang D, Liu S, Li Z, Wang R. Global, regional and national burden of gastroesophageal reflux disease, 1990-2019: update from the GBD 2019 study. Ann Med. 2022 Dec;54(1):1372-1384. doi: 10.1080/07853890.2022.2074535. PMID 35579516
- [Result] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT06928350/Prot_SAP_ICF_000.pdf